CLINICAL TRIAL: NCT03563300
Title: Gluten-related Disorders in Patients Affected With Familial Mediterranean Fever
Brief Title: Gluten-related Disorders in Familial Mediterranean Fever Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Pasquale Mansueto, Clinical Professor, University of Palermo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: ACPM21
Record Dates: First submitted 2018-05-24; First posted 2018-06-20 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Not-celiac Wheat Sensitivity (NCWS); Familial Mediterranean Fever (FMF)
MeSH Terms: conditions — Familial Mediterranean Fever | interventions — Flour

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wheat flour (Active Comparator): Wheat flour will be administered blindly versus placebo for 7 days
  Interventions: Other: Wheat flour
- Rice flour (Placebo Comparator): Placebo will be administered blindly versus wheat flour for 7 days
  Interventions: Other: Placebo Comparator

INTERVENTIONS:
Other: Wheat flour — Wheat flour will be administered once daily for 7 days
  Other Names: Active Comparator
  Arms: Wheat flour
Other: Placebo Comparator — Placebo will be administered blindly versus wheat flour for 7 days
  Other Names: Rice flour
  Arms: Rice flour

SUMMARY:
It is known that the gluten-containing grains can be responsible for human diseases related to gluten exposure. These forms of gluten intolerance represent a heterogeneous set of conditions, including celiac disease (CD), wheat allergy (WA) and not celiac gluten sensitivity (NCGS), that combined seems to affect about 5-10% of the general population. NCGS is the most recent gluten-related disease, characterized by intestinal and extra-intestinal symptoms related to the ingestion of gluten-containing food, in subjects in whom either celiac disease or wheat allergy previously has been excluded. However, as it is not known what component of the cereals causes the symptoms in NCGS patients, the investigators prefer the label of "Not-celiac wheat sensitivity" (NCWS). Typically, the NCWS diagnosis is made by exclusion. Furthermore, similarly to CD, the investigators had demonstrated that NCWS may be associated with other autoimmune disease (i.e. Hashimoto's thyroiditis). Among these autoimmune conditions, in our daily out clinic work, the investigators have observed an association between self-reported NCWS and Familial Mediterranean Fever (FMF). Our preliminary observational data indicate that some FMF patients relate their symptoms (especially gastrointestinal) to gluten assumption, then excluding it from diet and using gluten-free products, with partial remission of gastrointestinal symptoms. Therefore, FMF and NCGS share some clinical features, such as abdominal pain, diarrhea, arthralgia and arthritis, and tend to be commonly associated with other inflammatory and autoimmune diseases. This study has 2 major aims: 1.To evaluate the real relationship between the wheat ingestion and the gastrointestinal manifestations presented by FMF patients, self-reporting a NCWS. 2. To identify possible immunologic markers that may explain the mechanism underling FMF abdominal attack and wheat ingestion.

DETAILED DESCRIPTION:
It is known that the gluten-containing grains can be responsible for human diseases related to gluten exposure. These forms of gluten intolerance represent a heterogeneous set of conditions, including celiac disease (CD), wheat allergy (WA) and not celiac gluten sensitivity (NCGS), that combined seems to affect about 5-10% of the general population. NCGS is the most recent gluten-related disease. It is characterized by intestinal (i.e. irritable bowel syndrome, bloating, dyspepsia) and extra-intestinal symptoms (i.e. fatigue, headache, numbness, mental confusion) related to the ingestion of gluten-containing food, in subjects in whom either celiac disease or wheat allergy previously has been excluded. However, as it is not known what component of the cereals causes the symptoms in NCGS patients, the investigators prefer the label of "Not-celiac wheat sensitivity" (NCWS). Typically, the NCWS diagnosis is made by exclusion. In fact, in previous studies the investigators showed that patients self-reporting gastrointestinal symptoms related to wheat ingestion, could suffer not only from CD or WA, but from small intestinal bacterial overgrowth or inflammatory bowel diseases also. Furthermore, similarly to CD, the investigators had demonstrated that NCWS may be associated with other autoimmune disease (i.e. Hashimoto's thyroiditis). Among these autoimmune conditions, in our daily out clinic work, the investigators have observed an association between self-reported NCWS and Familial Mediterranean Fever (FMF). Familial Mediterranean fever (FMF) is the most frequent hereditary autoinflammatory disease, characterized by self-limited recurrent attacks of fever and serositis, resulting in pain in the abdomen, chest, joints and muscles. FMF is caused by mutations in MEFV gene, which encodes pyrin. Pyrin is implicated in a complex interplay with proteins involved in Toll-like receptor (TLR) signalling, PYD superfamily and procaspase-1 activation, suggesting a controlling role in inflammatory response. Abdominal pain is the most frequent symptom encountered in FMF; 95% of patients report this as the main symptom during at least some of their fever episodes, while 50% cite such an 'abdominal attack' as the first symptom of their disease. Presentation of a typical abdominal attack will resemble that of 'acute abdomen'. Onset is sudden and acute, leading to rapid development of symptoms within 1-2 hours. The abdominal pain is usually diffuse throughout the entire abdomen, although in some cases it may be localized; it may be very severe in intensity. This may be accompanied by any bowel activity, ranging from constipation (most often) to diarrhoea. The intensity of symptoms and signs of an inflammatory attack in FMF will decrease spontaneously after 12-24 hours, and usually, the attack resolves over the following 48 hours. Thus, after about 3 days the patient will be symptom-free again. Furthermore, so-called "incomplete" abdominal attacks may occur in FMF patients. These differ from 'typical' abdominal attacks in 1 or 2 features, which may include absence of fever, absence of 'true' peritonitis and/or localisation of the abdominal pain to a single specific abdominal area, minimal change in acute phase parameters. It may be difficult to differentiate an 'incomplete' abdominal attack from other causes of abdominal pain, mainly because of its atypical presentation. Our preliminary observational data indicate that some FMF patients relate their symptoms (especially gastrointestinal) to gluten assumption, then excluding it from diet and using gluten-free products, with partial remission of gastrointestinal symptoms. Therefore, FMF and NCGS share some clinical features, such as abdominal pain, diarrhea, arthralgia and arthritis, and tend to be commonly associated with other inflammatory and autoimmune diseases. However, to our knowledge, a relationship between FMF and NCGS has not been previously investigated. This study has 2 major aims: 1.To evaluate the real relationship between the wheat ingestion and the gastrointestinal manifestations presented by FMF patients, self-reporting a NCWS. The study will be done after a period of gluten-free diet, administering wheat flour or placebo for 15 days. 2. To identify possible immunologic markers (histological features, expression of cytokines and other constitutive mucosal proteins from peripheral blood mononuclear cells and mucosal lymphocytes) that may explain the mechanism underling FMF abdominal attack and wheat ingestion.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, both genders, with age between 18-65 years, affected with FMF, diagnosed according to clinical criteria designed by Livneh et al ("Tel-Hashomer" criteria), self-reporting a relationship between their symptoms (especially gastrointestinal) and gluten assumption, improving on a gluten-free diet and worsen on a gluten containing diet
* Patients testing negative for celiac disease (anti-tTG and EMA negative, and with biopsy Marsh 0-1) and wheat allergy (serum specific IgE for wheat negative)

Exclusion Criteria:

* Subjects diagnosed with celiac disease (positive anti-tTG and/or EMA, and positive histology, with Marsh 2 or above);
* Subjects diagnosed with wheat allergy (positive serum specific IgE for wheat)
* Subjects with Inflammatory Bowel Diseases (Crohn's disease or ulcerative colitis)
* Subjects with Helicobacter pylori infection and other gastrointestinal infection
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Fibromyalgia symptoms evaluation | Change from baseline at 1 week
  Fibromyalgia symptoms of patients, evaluated by the International Severity Scoring System for Familial Mediterranean Fever (ISSF), will be scored before and after 1 week of wheat (or placebo) ingestion
Gastrointestinal symptoms evaluation | Change from baseline at 1 week
  Gastrointestinal symptoms of patients, evaluated by the Gastrointestinal Symptom Rating Scale (GSRS), will be scored before and after 1 week of wheat (or placebo) ingestion

SECONDARY OUTCOMES:
Leukocytes cell surface antigens expression | Change from baseline at 1 week
  There will be evaluated some leukocytes cell surface antigens expression, i.e. CD45, CD56, CD117, NKp44, CD3, CD19, and CD14, from peripheral blood mononuclear cells and rectal mucosal lymphocytes before and after 1 week of wheat (or placebo) ingestion
Cytokines production | Change from baseline at 1 week
  There will be evaluated some cytokines production, i.e. IFN-γ, TNF-α, IL-22, IL-17, and T-bet, from peripheral blood mononuclear cells and rectal mucosal lymphocytes before and after 1 week of wheat (or placebo) ingestion

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Carroccio, PhD, Principal Investigator — University of Palermo
Locations (2):
- Italy (2):
  - Department of Internal Medicine, Giovanni Paolo II Hospital of Sciacca, Sciacca, Agrigento
  - Department of Internal Medicine, University Hospital of Palermo, Palermo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Carroccio A, Mansueto P, Iacono G, Soresi M, D'Alcamo A, Cavataio F, Brusca I, Florena AM, Ambrosiano G, Seidita A, Pirrone G, Rini GB. Non-celiac wheat sensitivity diagnosed by double-blind placebo-controlled challenge: exploring a new clinical entity. Am J Gastroenterol. 2012 Dec;107(12):1898-906; quiz 1907. doi: 10.1038/ajg.2012.236. Epub 2012 Jul 24. PMID 22825366
- [Result] Carroccio A, Mansueto P, D'Alcamo A, Iacono G. Non-celiac wheat sensitivity as an allergic condition: personal experience and narrative review. Am J Gastroenterol. 2013 Dec;108(12):1845-52; quiz 1853. doi: 10.1038/ajg.2013.353. Epub 2013 Nov 5. PMID 24169272
- [Result] Carroccio A, Rini G, Mansueto P. Non-celiac wheat sensitivity is a more appropriate label than non-celiac gluten sensitivity. Gastroenterology. 2014 Jan;146(1):320-1. doi: 10.1053/j.gastro.2013.08.061. Epub 2013 Nov 22. No abstract available. PMID 24275240
- [Result] Mansueto P, Seidita A, D'Alcamo A, Carroccio A. Non-celiac gluten sensitivity: literature review. J Am Coll Nutr. 2014;33(1):39-54. doi: 10.1080/07315724.2014.869996. PMID 24533607
- [Result] Carroccio A, D'Alcamo A, Cavataio F, Soresi M, Seidita A, Sciume C, Geraci G, Iacono G, Mansueto P. High Proportions of People With Nonceliac Wheat Sensitivity Have Autoimmune Disease or Antinuclear Antibodies. Gastroenterology. 2015 Sep;149(3):596-603.e1. doi: 10.1053/j.gastro.2015.05.040. Epub 2015 May 27. PMID 26026392
- [Result] Di Liberto D, Mansueto P, D'Alcamo A, Lo Pizzo M, Lo Presti E, Geraci G, Fayer F, Guggino G, Iacono G, Dieli F, Carroccio A. Predominance of Type 1 Innate Lymphoid Cells in the Rectal Mucosa of Patients With Non-Celiac Wheat Sensitivity: Reversal After a Wheat-Free Diet. Clin Transl Gastroenterol. 2016 Jul 7;7(7):e178. doi: 10.1038/ctg.2016.35. PMID 27388423
- [Result] Demirkaya E, Acikel C, Hashkes P, Gattorno M, Gul A, Ozdogan H, Turker T, Karadag O, Livneh A, Ben-Chetrit E, Ozen S; FMF Arthritis Vasculitis and Orphan disease Research in pediatric rheumatology (FAVOR). Development and initial validation of international severity scoring system for familial Mediterranean fever (ISSF). Ann Rheum Dis. 2016 Jun;75(6):1051-6. doi: 10.1136/annrheumdis-2015-208671. Epub 2016 Jan 28. PMID 26823530
- [Result] Svedlund J, Sjodin I, Dotevall G. GSRS--a clinical rating scale for gastrointestinal symptoms in patients with irritable bowel syndrome and peptic ulcer disease. Dig Dis Sci. 1988 Feb;33(2):129-34. doi: 10.1007/BF01535722. PMID 3123181